CLINICAL TRIAL: NCT06251206
Title: Impact of Early Multimodal ADL Education on Outcomes Post Distal Radius Fracture Open Reduction Internal Fixation Surgery
Brief Title: Impact of Early ADL Education on Outcomes Post DRF ORIF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Sarah Doerrer, Assistant Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCR235402
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Distal Radius Fractures
Keywords: Activities of Daily Living; Postsurgical Patient Education
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADL/Postoperative Instruction (Experimental): Participants in the experimental group will watch a video instructing them on early ADL participation after DRF fracture treated by ORIF and postoperative care. Participants in the experimental group will also receive a handout on ADL participation and postoperative care with a QR code to the video.
  Interventions: Behavioral: ADL/Postoperative Instruction; Behavioral: Postoperative Instruction
- Postoperative Instruction (Active Comparator): Participants in the control group will watch a video instructing them on postoperative care. Participants in the control group will receive a handout on postoperative care with a QR code to the video.
  Interventions: Behavioral: Postoperative Instruction

INTERVENTIONS:
Behavioral: ADL/Postoperative Instruction — This is an education video which includes demonstration of simple ADL tasks that the participant can do at home after surgery. Handout includes the same information and a QR code to watch the video.
  Arms: ADL/Postoperative Instruction
Behavioral: Postoperative Instruction — This is an education video that only includes the postoperative instructions. Handout includes the same information and a QR code to watch the video.

SUMMARY:
This study is a randomized controlled trial (RCT). This RCT which will study the effect of performing daily activities early after a distal radius fracture being treated with surgical intervention of open reduction and internal fixation. This study will have two groups. The experimental group will watch a video and be given a handout on how to perform daily activities with the hand of the injured wrist while recovering from surgery and postoperative instructions. The control group will watch a video on wound care and be given a handout on postoperative instructions. Outcome measures will be taken at initial evaluation between 1-2 weeks post surgery, at 5-7 weeks post surgery, at 8-10 weeks, and at 12-14 weeks. Outcome measures will include the Michigan Wrist Evaluation, Visual Analog Pain Scale, Tampa Scale of Kinesiophobia-11 Scale, finger mobility testing, grip and pinch strength, and the 9 hole peg test to test fine motor coordination. Outcome measure scores will be compared between groups using a t-test statistical test. Outcome measure scores will also be tested within groups using a paired t-test.

DETAILED DESCRIPTION:
1. The surgeon will recruit patients who have had surgery for a distal radius fracture with open reduction and internal fixation and have met inclusion and exclusion criteria utilizing a recruitment statement.
2. If the patient is interested in participating in the study, the surgeon will obtain informed consent and email a copy of the informed consent form to the patient.
3. Once informed consent is obtained, the surgeon will ask the front desk to give him an envelop which will include a letter with either the word control or experimental group on it.
4. Once the surgeon reads the letter, the subject will receive either the standard of care video and handout (control) or the intervention video and handout (experimental).
5. If the subject receives the intervention then the surgeon will play the intervention video in the office and review with the subject the educational handout. The handout will be given to the subject to take home which includes a QR code to the educational video.

If the subject is in the control group then the surgeon will play the standard of care (postoperative care) video in the office and review with the subject the postoperative care handout. The handout will be given to the subject to take home which includes a QR code to the video.

The following data collection procedures will occur with the subjects

The surgeon will collect data from all subjects at 1-2 weeks post surgery and data collection will include: age, gender, race, hand dominance, side injured, fracture severity, workers comp status, comorbidities, smoker status, work status, and household assistance. The hand surgeon will also collect data from the subjects on their current level of function, pain, and fear of moving their injured limb.

At 5-7 weeks the surgeon will collect data from all subjects on their current level of function, pain, fear of moving their injured limb. The surgeon will also measure finger motion.

At 8-10 weeks the surgeon will collect data from all subjects on their current level of function, pain, fear of moving their injured limb. The surgeon will also measure finger motion, grip, pinch strength and fine motor coordination.

At 12-14 the surgeon will collect data from all subjects on their current level of function, pain, fear of moving their injured limb. The surgeon will also measure finger motion, grip, pinch strength and fine motor coordination.

All subjects will be followed for 14 weeks. If the patient receives a referral for hand therapy it will be noted in the record. It will also be noted in the record if subject experiences any complication such as median nerve compression, tendonitis, or complex regional pain syndrome.

The outcome measures that will be used with both the control and experimental groups and at each time point that the data will be collected. All outcome measures will be uploaded onto RedCap. Subjects will use a tablet to fill out all questionnaires (Michigan Hand Evaluation, Visual Analog Scale, Tampa Scale of Kinesiophobia-11) while in the office or forms will be emailed through RedCap and scores will be uploaded into the RedCap database. All clinical tests (grip and pinch testing, distance from distal palmar crease, 9 hole peg test) will be recorded in RedCap. Demographic information will either be collected on the tablet in RedCap.

ELIGIBILITY:
Inclusion Criteria:

English Speaking DRF treated with ORIF Individuals 18 years of age or older 2 weeks or less post ORIF for DRF

Exclusion Criteria:

Individuals with pre-existing neurological coniditons affecting the upper limb Individuals with congnitive deficits that would limit the ability to correctly report information on outcome measures Individuals with psychological deficits which would limit the ability to correctly report information on outcome measures Individuals with multiple injuries to the affected upper limb Individuals with multiple injuries to both upper limbs Prior distal radius fracture involving the same wrist Individuals receiving hand therapy for another injury at enrollment into study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Michigan Hand Questionnaire | baseline, 5-7 weeks, 8-10 weeks, 12-14 weeks
  Patient reported outcome measure for function

SECONDARY OUTCOMES:
Visual Analog Scale | baseline, 5-7 weeks, 8-10 weeks, 12-14 weeks
  patient reported outcome measure for pain intensity
Tampa Scale of Kinesiophobia | baseline, 5-7 weeks, 8-10 weeks, 12-14 weeks
  patient reported outcome measure for fear of movement
Range of Motion of digits | 5-7 weeks, 8-10 weeks, 12-14 weeks
  distance from digits to distal palmar crease in cm
Grip and Pinch Strength | 8-10 weeks, 12-14 weeks
  Jamar grip gauge testing and pinchmeter gauge testing for strength
9 hole peg test | 8-10 weeks, 12-14 weeks
  fine motor coordination/sensorimotor test

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Facilities Associates, Washington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No